CLINICAL TRIAL: NCT04003493
Title: LifE Style, Nutrition and Oral Health in Care Givers)
Brief Title: LifE Style, Nutrition and Oral Health in Care Givers (LENTO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Collaborators: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LENTO
Record Dates: First submitted 2019-06-25; First posted 2019-07-01 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Nutrition Disorders in Old Age; Caries,Dental; Dentures; Oral Mucositis; Tooth Diseases; Plaque, Dental; Gingival Diseases
Keywords: Nutrition; Oral health; Care givers; Home care clients; Quality of life
MeSH Terms: conditions — Dental Caries; Stomatitis; Tooth Diseases; Dental Plaque; Gingival Diseases | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention group of nutrition (Experimental): On the basis of a blood test, Mini Nutritional Assessment, food diary and nutritional anamnesis, the nutritionist developed a plan for individualised nutritional care and discussed with the caregivers. If the caregivers seemed unable to increase the energy and/or protein of their diet, daily complementary dietary drinks were recommended to them. The participants were re-examined six months after the baseline interviews to evaluate the effectiveness of the interventions.
  Interventions: Other: Nutrition and oral health intervention
- Control group of nutrition (No Intervention): The control group has the same examinations as the intervention group, they do not get dietary counseling.
- Intervention group of oral health (Experimental): After the dental hygienist interview and oral health examination, the caregivers in need were targeted for oral health intervention. The intervention included individualised instructions on either dental hygiene, denture hygiene, cleaning of the oral mucosa or for dry mouth. The participants were re-examined six months after the baseline interviews to evaluate the effectiveness of the interventions.
  Interventions: Other: Nutrition and oral health intervention
- Control group of oral health (No Intervention): The control group has the same examinations as the intervention group, they do not get oral health counseling.

INTERVENTIONS:
Other: Nutrition and oral health intervention — The interventions included individualised nutrition and oral health care.
  Arms: Intervention group of nutrition; Intervention group of oral health

SUMMARY:
The LENTO study sample includes the caregivers and their clients living in eastern Finland. The aims of this study are

1. to study the nutritional status, oral health, coping, functional capacity and quality of life
2. to find out how individual nutrition and oral health counseling received for caregivers affect on the nutritional status and oral health of caregivers and their clients
3. develop an operating model to maintain good nutrition and oral health.

DETAILED DESCRIPTION:
In Finland, the aim is to reduce the institutional care of older people and caring them in their own homes. The goal of shifting the focus of services to open services is difficult to implement if the health of the caregivers is inadequate. In order to achieve this goal, it is important to influence the health and performance of caregivers. Information is needed to support this, among others, about how the nutrition and oral health of caregivers can be promoted and to what extent this affects the performance and quality of life of their clients. A randomly of 220 caregivers over 65 years old and their clients is selected for this study. The caregivers are randomized to either treatment or control groups. At the beginning of the study is estimated the nutritional status and oral health of the caregivers. Based on the results, the nutritionist and dental hygienist give individual advice to optimize the nutrition and oral health of the caregivers in the intervention group. After six months, the same measurements are made as at the beginning of the study. Monitoring measurements will be made one year after the start of the intervention. The results of this project provide information on the health, well-being, and ability to the function of the caregivers. Based on the results, is developed an operating model that is intended to be wide as use as possible. Improving the nutrition and oral health of caregivers has a significant impact on their own and their clients health and well-being as well as the long-term care costs presumably.

ELIGIBILITY:
Inclusion Criteria:

* caregivers who have a caregiver´s contract valid on 1 January 2019
* care recipients living at home

Exclusion Criteria:

* in terminal care

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 250 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Nutritional status | Baseline and 6 months and (12 months follow-up visit)
  Change in MNA scores
Albumin | Baseline and 6 months and (12 months follow-up visit)
  Change in plasma albumin concentration
Prealbumin | Baseline and 6 months and (12 months follow-up visit)
  Change in plasma prealbumin concentration
Body mass index (kg/m2) | Baseline and 6 months and (12 months follow-up visit)
  Change in BMI
Hand grip strength | Baseline and 6 months and (12 months follow-up visit)
  Change in had grip strength of boot hands
Number and location of teeth | Baseline and 6 months and (12 months follow-up visit)
  Change in number and location of teeth
Type and location of removable dental prosthesis | Baseline and 6 months and (12 months follow-up visit)
  Change in type and location of removable dental prosthesis
Oral mucosa | Baseline and 6 months and (12 months follow-up visit)
  Change in oral mucosa
Condition of teeth | Baseline and 6 months and (12 months follow-up visit)
  Change in condition of teeth
Presence of plaque | Baseline and 6 months and (12 months follow-up visit)
  Change in presence of plaque
Gingival bleeding and measurement of periodontal pockets | Baseline and 6 months and (12 months follow-up visit)
  Change in gingival bleeding and measurement of periodontal pockets
Dental and denture hygiene | Baseline and 6 months and (12 months follow-up visit)
  Change dental and denture hygiene
Subjective feeling of dry mouth and pain in mouth | Baseline and 6 months and (12 months follow-up visit)
  Change in subjective feeling of dry mouth and pain in mouth

SECONDARY OUTCOMES:
Activities of Daily Living | Baseline and 6 months and (12 months follow-up visit)
  Change in Activities of Daily Living (ADL) scores
Instrumental Activities of Daily Living | Baseline and 6 months and (12 months follow-up visit)
  Change in Instrumental Activities of Daily Living (IADL) scores
Quality of Life (WHOQOL) -bref scores | Baseline and 6 months and (12 months follow-up visit)
  Change in quality of Life (WHOQOL) -bref scores
Depression | Baseline and 6 months and (12 months follow-up visit)
  Change in Geriatric Depression Scale (GDS)-15 scores
Cognition | Baseline and 6 months and (12 months follow-up visit)
  Change in Mini Mental State Examination (MMSE) scores
Sense of coherence | Baseline and 6 months and (12 months follow-up visit)
  Change in sense of coherence (SOC) scores
Morbidity | Baseline
  Functional Comorbidity Index (FCI) scores

CONTACTS AND LOCATIONS:
Overall Officials: Ursula o Schwab, PhD, Study Director — Study Principal Inverstigator, professor; Liisa o Suominen, PhD, Principal Investigator — Study Principal Inverstigator, professor; Tarja o Välimäki, PhD, Principal Investigator — Study Principal Inverstigator, adjuct professor; Irma o Nykänen, PhD, Principal Investigator — Study Principal Investigator, adjuct professor
Locations (1):
- University of Eastern Finland, Kuopio, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Annina S, Irma N, Tarja V, Sohvi K, Roosa-Maria S, Ursula S, Suominen AL. The Effect of an Individually Tailored Oral Health Intervention on Dental Plaque and Caries Among Family Caregivers and Their Care Recipients. Gerodontology. 2025 Dec;42(4):495-506. doi: 10.1111/ger.12814. Epub 2025 Mar 25. PMID 40129259
- [Derived] Koponen S, Nykanen I, Savela RM, Valimaki T, Suominen AL, Schwab U. Underweight, overweight, and weight change in older family caregivers and their care recipients: longitudinal evidence from a randomized controlled trial. Front Aging. 2024 Aug 15;5:1376825. doi: 10.3389/fragi.2024.1376825. eCollection 2024. PMID 39211745
- [Derived] Koponen S, Nykanen I, Savela RM, Valimaki T, Suominen AL, Schwab U. Family caregivers' better nutritional status is associated with care recipients' better nutritional status. Clin Nutr ESPEN. 2024 Aug;62:199-205. doi: 10.1016/j.clnesp.2024.05.016. Epub 2024 May 28. PMID 38901942
- [Derived] Razzaq S, Nykanen I, Valimaki T, Koponen S, Savela RM, Schwab U, Suominen AL. Use of oral health care services by family caregivers and care recipients: the LENTO intervention. Acta Odontol Scand. 2024 May 22;83:317-326. doi: 10.2340/aos.v83.40687. PMID 38775632
- [Derived] Koponen S, Nykanen I, Savela RM, Valimaki T, Suominen AL, Schwab U. Depressive symptoms, low-grade inflammation, and poor oral health prevents the success of nutritional guidance in older caregivers. Clin Nutr ESPEN. 2023 Oct;57:39-47. doi: 10.1016/j.clnesp.2023.06.018. Epub 2023 Jun 22. PMID 37739684
- [Derived] Koponen S, Nykanen I, Savela RM, Valimaki T, Suominen AL, Schwab U. Individually tailored nutritional guidance improved dietary intake of older family caregivers: a randomized controlled trial. Eur J Nutr. 2022 Oct;61(7):3585-3596. doi: 10.1007/s00394-022-02908-w. Epub 2022 May 27. PMID 35622137
- [Derived] Nykanen I, Valimaki T, Suominen L, Schwab U. Optimizing nutrition and oral health for caregivers-intervention protocol. Trials. 2021 Sep 15;22(1):625. doi: 10.1186/s13063-021-05589-8. PMID 34526071